CLINICAL TRIAL: NCT05456334
Title: New Treatments for Actinic Keratoses of the Scalp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kirsi Isoherranen, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-001268-12
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Photodamaged Skin; Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Lasers, Dye

STUDY DESIGN:
Intervention Model Description: half-side comparative randomized controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pulsed dye laser-mediated photodynamic therapy (Experimental): After curretage light-sensitizer (methyl aminolaevulinate cream) was applied on the lesions and covered with an occlusive plastic foil for 2-3-h incubation. Then a local lidocaine anaesthetic spray was applied. The lesions were illuminated with 30% overlapping pulsed laser double-stacked pulses (, energy 7 J/cm2, spot size 7 mm, pulse duration 10 ms, wavelength 595 nm and dynamic cooling 2/3).
  Interventions: Device: Pulsed-dye laser; Drug: Metvix cream
- Conventional photodynamic therapy (Active Comparator): After curretage a light-sensitizer (methyl aminolaevulinate cream) was applied on the lesions and covered with an occlusive plastic foil for 2-3-h incubation. Then a local lidocaine anaesthetic spray was applied. The lesions were illuminated with a red LED light for 7-8 min (exposure 75 J/cm2, wavelength 630 nm).
  Interventions: Drug: Metvix cream
- Ablative fractional laser- mediated daylight photodynamic therapy (Experimental): After curretage lidocaine anaesthetic spray was applied on the whole treatment area. Lesions were treated with an ablative fractional CO2-laser (19 W, Dot mode, spacing 1000 µm, stack 3, scanning dwell time 1800 µs, repeat 0.5 s). A thin layer of light sensitizer (methyl aminolaevulinate cream) was applied on the treatment area. The patients were asked to move outdoors (temperature >10C, no rain, June-August) or to our adPDT-room (IndoorLux®, wavelength 350-750 nm, 15-25 000 lux) within 30 minutes, for the 2h-illumination.
  Interventions: Device: Fractional CO2-laser; Drug: Metvix cream
- Daylight photodynamic therapy (Active Comparator): After curretage lidocaine anaesthetic spray was applied on the whole treatment area. A thin layer of light sensitizer (methyl aminolaevulinate cream) was applied on the treatment area. The patients were asked to move outdoors (temperature >10C, no rain, June-August) or to our adPDT-room (IndoorLux®, wavelength 350-750 nm, 15-25 000 lux) within 30 minutes, for the 2h-illumination.
  Interventions: Drug: Metvix cream

INTERVENTIONS:
Device: Pulsed-dye laser — Comparance of pulsed-dye laser-mediated and conventional photodynamic therapy in a split-head design
  Arms: Pulsed dye laser-mediated photodynamic therapy
Device: Fractional CO2-laser — Comparance of fractional CO2-laser-mediated or plain daylight photodynamic therapy in a split-head design
  Arms: Ablative fractional laser- mediated daylight photodynamic therapy
Drug: Metvix cream — Metvix-cream was used for photodynamic therapy in all experimental arms

SUMMARY:
This blinded controlled 2-year study on 120 patients with 2 or more actinic keratoses, compare the efficacy and tolerability of pulsed dye-laser- mediated photodynamic therapy compared to conventional photodynamic therapy and fractional-laser assisted daylight photodynamic therapy compared to daylight photodynamic therapy.

DETAILED DESCRIPTION:
Actinic keratoses are premalign skin lesions with increasing prevalence, causing a rising burden on the health care system. In this blinded controlled study we assess the efficacy of pulsed dye-laser- mediated photodynamic therapy compared to conventional photodynamic therapy and fractional-laser assisted daylight photodynamic therapy to daylight photodynamic therapy. It is a prospective, randomized and blinded split-head comparative study during the years 2016- 2024. 120 patients are recruited based on referral or from patients attending the clinic, with 2 or more actinic keratoses on the head, 60 to the pulsed dye-laser study and 60 to the fractional laser study. Follow-up appointments are 6 months, 1 year and 2 years post treatment. Patient reported maximal pain during treatment is documented.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 AKs located on both sides of the head (either the scalp, forehead, temples, or cheeks)

Exclusion Criteria:

* pigmented AKs, in situ-carcinomas, skin cancers, psoriasis or eczema on the treatment area

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient complete (%, P) or partial clearance (%, P) | 2 year
  All actinic keratoses on the particular treatment area cleared, or 75% of lesions on treatment area cleared
Lesion-specific clearance (%, P) | 2 year
  Proportion of lesions that completely healed, partially healed or not healed in the particular treatment

SECONDARY OUTCOMES:
Patient reported pain | 1 day
  Maximal pain during treatment on the Numerical Rating Scale (0-10)

IPD SHARING:
Plan to Share IPD: No